CLINICAL TRIAL: NCT04507165
Title: The Effect of Opioid-free Anesthesia on Postoperative Analgesia-related Adverse Reactions in Lung Resection With Video-assisted Thoracoscopic Access: a Randomized Double-blind Controlled Study
Brief Title: Opioid-free Anesthesia in VATS Lung Resection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Yi Feng, MD, Chief of the Anesthesiology Department, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020PHB031
Record Dates: First submitted 2020-07-31; First posted 2020-08-11 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Opioid Free Anesthesia
Keywords: Opioid Free Anesthesia; Video-assisted Thoracoscopic Surgery
MeSH Terms: interventions — Nerve Block

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- opioid-free general anesthesia (Experimental): under opioid-free general anesthesia
  Interventions: Procedure: Paravertebral block+Anterior serratus plane block; Drug: opioid free anesthesia
- opioid based general anesthesia (Active Comparator): under opioid based general anesthesia
  Interventions: Procedure: Paravertebral block+Anterior serratus plane block; Drug: opioid based anesthesia

INTERVENTIONS:
Procedure: Paravertebral block+Anterior serratus plane block — Paravertebral block will be performed at T3 and T7 level on the surgical side using out-of-plane approach under ultrasound-guided, with 0.5% ropivacaine 10ml at each injection site. Anterior serratus plane block will be performed at the 4th rib level on the surgical side under ultrasound-guided, with 0.5% ropivacaine 15ml. The blocking range is measured by "ice cube" method 15 minutes after the procedure.
  Other Names: nerve block
Drug: opioid free anesthesia — Anesthesia induction: Dexmedetomidine 1µg/kg (intravenous infusion within 10min), propofol 1.5-2mg/kg (intravenous bolus), lidocaine 1.5-2mg/kg (intravenous bolus), cisatracurium besylate 0.15-0.3mg/kg (intravenous bolus before tracheal intubation), methylprednisolone 40mg (intravenous bolus), esmolol 1mg/kg (intravenous bolus), and 0.5% tetracaine 5ml for surface anesthesia of the throat.
  Maintenance of anesthesia: Continuous infusion of propofol and dexmedetomidine [0.4μg/(kg.h)]. The infusion rate of propofol was adjusted according to bispectral index value. Cisatracurium besylate was given as needed. Flurbiprofen 50mg was given intravenously before the skin incision and suture respectively.
  Remedy: If blood pressure rises (more than 30% of the mean arterial pressure after induction), and heart rate increases (more than 30% of heart rate after induction) during skin incision, lidocaine 1.5mg/kg will be given intravenously and then be continuously infused at a rate of 1.5mg/(kg.h).
  Other Names: OFA
  Arms: opioid-free general anesthesia
Drug: opioid based anesthesia — Anesthesia induction: Propofol 1.5-2mg/kg (intravenous bolus), sufentanil 0.3μg/kg (intravenous bolus), cisatracurium besylate 0.15-0.3mg/kg (intravenous bolus before tracheal intubation), methylprednisolone 40mg (intravenous bolus), esmolol 1mg/kg (intravenous bolus).
  Maintenance of anesthesia: Continuous infusion of propofol and remifentanil. The infusion rate of propofol was adjusted according to BIS value. The infusion rate of remifentanil was 0.1-0.5µg/(kg.min) and adjusted according to the change of heart rate and blood pressure. Cisatracurium besylate was given as needed. Sufentanil 0.1μg/kg and flurbiprofen 50mg were given intravenously before the skin incision and suture respectively.
  Other Names: Standard anesthesia
  Arms: opioid based general anesthesia

SUMMARY:
A comparison of incidences of postoperative opioid-related adverse effects and recovery parameters in patients undergoing video-assisted thoracoscopic surgery (VATS) lung resection receiving opioid or opioid-free general anesthesia (OFA).

DETAILED DESCRIPTION:
Video-assisted thoracoscopic surgery (VATS) lung resection is traditionally performed under general anesthesia with opioid-based analgesia. It is associated with higher incidences of respiratory depression, hypotension, postoperative nausea and vomiting (PONV), dizziness, constipation and urinary retention, and more severe acute postoperative pain.

The purpose of our study is to compare the opioid-free general anesthesia with the opioid-based general anesthesia with respect to the primary outcome measures of the total incidence of opioid-related adverse effects (including respiratory depression, hypotension, PONV and dizziness) and secondary outcome measures of incidence of intraoperative and postoperative cardiovascular complications, pain relief, analgesic requirement , and other postoperative recovery parameters [e.g. duration of tracheal extubation, departing from post-anaesthesia care unit (PACU), exhaust, defecation, and stay in hospital postoperatively].

ELIGIBILITY:
Inclusion Criteria:

* Undergoing VATS lung resection.
* American Society of Anesthesiologists (ASA) physical status I-II.
* Agreed to participate in the trial.

Exclusion Criteria:

* Pregnant women
* ASA phase III or above.
* Undergoing emergency surgery.
* Planning for thoracotomy.
* Adults protected by law (under judicial protection, guardianship or supervision), people who deprived of their liberty.
* Patients who have received general anesthesia.
* Atrioventricular block, sinus node block or intraventricular block.
* Sinus bradycardia (heart rate is less than 60 beats/min).
* Preoperative hypotension (systolic blood pressure is less than 90mmHg)
* Combined with urolithiasis, Meniere syndrome, and vertebral artery stenosis
* Combined with cerebrovascular disease.
* Contraindication to NSAIDs drug.
* Allergic to anesthetics.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Total incidence of opioid-related adverse effects of 2 hours, 4 hours, 6 hours, 24 hours and 48 hours postoperation | 2 hours, 4 hours, 6 hours, 24 hours and 48 hours postoperation
  The total incidence refers to the sum of the incidence of opioid-related adverse effects at 2h, 4h, 6h, 24h and 48h postoperationOpioid-related adverse effects here including respiratory depression, hypotension, PONV and dizziness.

SECONDARY OUTCOMES:
Incidence of intraoperative cardiovascular complications | During the operation
  Including the incidence of arrhythmia, the probability of using hyperensor and hypotensor.
Incidence of postoperative cardiovascular complications | Up to 30 days postoperation
  Including the incidence of arrhythmia, the probability of using hypertensor and hypotensor.
Duration of tracheal intubation removing | Up to 2 hours postoperation
  From anesthetic discontinuance to tracheal extubation
Duration of departing from PACU | Up to 4 hours postoperation
  From tracheal extubation to Aldrete score>9. Aldrete score is the standard for departing from PACU which includes five contents to evaluate: activity, breath, blood pressure, state of consciousness and oxygen saturation by pulse oximetry (SpO2). 2 point in total for each content. 2 point refers to the best state, whereas 0 point refers to the worst state. When a patient's total score greater than 9 who will be transferred out of PACU.
Pain severity | 2 hours, 4 hours, 6 hours, 24 hours and 48 hours after tracheal extubation
  Using 0-10 numerical rating scale (NRS). The NRS score is ranged from 0 to 10. 0 means without pain. 1-3 means mild pain. 4-6 means moderate pain. 7-9 means severe pain. 10 means intense pain and can't bear.
Dosage of opioids | 2 hours, 4 hours, 6 hours, 24 hours and 48 hours after tracheal extubation
  Total dosage of opioids postoperation
Flatus time | Up to 48 hours postoperation
  From the operation finished to first-time exhaust
Defecation time | Up to 48 hours postoperation
  From the operation finished to first-time defecation
Postoperative duration of stay in hospital | 30 days postoperation
  The duration when patients stay in hospital after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Feng Yi, MD,PhD, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dinges HC, Otto S, Stay DK, Baumlein S, Waldmann S, Kranke P, Wulf HF, Eberhart LH. Side Effect Rates of Opioids in Equianalgesic Doses via Intravenous Patient-Controlled Analgesia: A Systematic Review and Network Meta-analysis. Anesth Analg. 2019 Oct;129(4):1153-1162. doi: 10.1213/ANE.0000000000003887. PMID 30418234
- [Background] Cozowicz C, Poeran J, Zubizarreta N, Liu J, Weinstein SM, Pichler L, Mazumdar M, Memtsoudis SG. Non-opioid analgesic modes of pain management are associated with reduced postoperative complications and resource utilisation: a retrospective study of obstructive sleep apnoea patients undergoing elective joint arthroplasty. Br J Anaesth. 2019 Jan;122(1):131-140. doi: 10.1016/j.bja.2018.08.027. Epub 2018 Oct 27. PMID 30579391
- [Background] Forget P. Opioid-free anaesthesia. Why and how? A contextual analysis. Anaesth Crit Care Pain Med. 2019 Apr;38(2):169-172. doi: 10.1016/j.accpm.2018.05.002. Epub 2018 Sep 13. PMID 29775728
- [Derived] Zhang R, Wu Y, Wang X, Zhang W, Feng Y. Efficacy of opioid-free anesthesia in reducing postoperative adverse events for thoracoscopic pulmonary surgery: a randomized controlled trial. BMC Anesthesiol. 2025 Dec 12;25(1):607. doi: 10.1186/s12871-025-03497-x. PMID 41388253